CLINICAL TRIAL: NCT00667121
Title: The Effect of Antidepressants and Gabapentin on Tamoxifen Pharmacokinetics: A Prospective Study
Brief Title: Tamoxifen in Women With Breast Cancer and in Women at High-Risk of Breast Cancer Who Are Receiving Venlafaxine, Citalopram, Escitalopram, Gabapentin, or Sertraline
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC0738; 07-006133 (Other: Mayo Clinic IRB); NCI-2011-00406 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Depression; Hot Flashes; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; breast cancer; hot flashes; depression
MeSH Terms: conditions — Breast Neoplasms; Depression; Hot Flashes | interventions — Citalopram; Escitalopram; Gabapentin; Sertraline; Tamoxifen; Venlafaxine Hydrochloride; Genetic Testing; Chromatography, High Pressure Liquid; Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: citalopram hydrobromide
Drug: escitalopram oxalate
Drug: gabapentin
Drug: sertraline hydrochloride
Drug: tamoxifen citrate
Drug: venlafaxine
Genetic: molecular genetic technique
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients receiving tamoxifen may help doctors learn more about the effects of other drugs on the level of tamoxifen in the blood.

PURPOSE: This clinical trial is studying levels of tamoxifen in the blood of women with breast cancer and in women at high risk of breast cancer who are receiving tamoxifen together with venlafaxine, citalopram, escitalopram, gabapentin, or sertraline.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine the changes in the plasma concentrations of the hydroxylated metabolite, 4-hydroxy tamoxifen, and endoxifen in women with known or at high risk for developing breast cancer who are receiving selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor therapy comprising venlafaxine, citalopram hydrobromide, escitalopram oxalate, gabapentin, or sertraline hydrochloride for the treatment of hot flashes, depression, or any other medically indicated condition.
* To evaluate whether genetic variants known to affect the activity of CYP2D6, SULT1A1, and other drug metabolizing enzymes (e.g., UGT's) involved in the biotransformation of tamoxifen citrate affect the plasma concentrations of the hydroxylated metabolites, 4-hydroxy tamoxifen and endoxifen.

OUTLINE: This is a multicenter study.

Patients receive oral tamoxifen citrate and concurrent selective serotonin reuptake inhibitor (SSRI)/serotonin-norepinephrine reuptake inhibitor (SNRI) therapy comprising oral venlafaxine, citalopram hydrobromide, escitalopram oxalate, sertraline hydrochloride, or gabapentin for 8-24 weeks. Treatment continues in the absence of disease progression.

Blood samples are obtained at baseline and after completion of study therapy. Samples are evaluated by pharmacokinetic analysis to determine the effects of SSRI/SNRI study drugs on plasma concentrations of tamoxifen and its metabolites. Plasma levels of tamoxifen citrate, N-desmethyl tamoxifen, 4-OH tamoxifen, and endoxifen are measured using reverse phase high performance liquid chromatography. Blood samples are also analyzed by CYP2D6 genotyping to test for CYP2D6 gene variation (i.e., *3, *4, *6, *10, *17, and *41) in genes that encode tamoxifen-metabolizing enzymes. Additional CYP2D6 alleles, including gene duplication and gene deletion (*5) are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed tamoxifen either for the prevention or treatment of non-invasive or invasive breast cancer.
* Tamoxifen use > 4 weeks without any breaks at a dose of 20 mg/day prior to registration
* to begin medical therapy with one of the following drugs: venlafaxine, citalopram, escitalopram, sertraline or gabapentin as determined by their physician
* Agree to continue tamoxifen during the proposed minimum study period of 8 weeks
* Willing to avoid known inhibitors of the CYP2D6 system for duration of study
* Ability to provide informed consent
* Willing to return to primary site of enrollment for follow-up
* Life expectancy >= 16 weeks
* Agree to provide a blood specimen at the time of pre-treatment (baseline) and at follow-up

Exclusion Criteria:

* Contraindication to the use of venlafaxine, citalopram, escitalopram, gabapentin or sertraline.
* Use of medications that are known to inhibit the CYP2D6 system within 3 weeks of registration. (see appendix II for list)
* Known to be a CYP2D6 poor metabolizer (defined as homozygous for one of the following CYP2D6 null alleles: *3, *4, *5, *6).

  * Note: CYP2D6 genotyping is not required prior to enrollment; however, CYP2D6 genotyping will be performed at baseline and the treating physician will be notified of the results: all genotypic CYP2D6 PM will be replaced

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENT CHARACTERISTICS:
  * Menopausal status not specified
  * Life expectancy ≥ 16 weeks
  * No contraindication for venlafaxine, citalopram hydrobromide, escitalopram oxalate, gabapentin, or sertraline hydrochloride
  PRIOR CONCURRENT THERAPY:
  * See Disease Characteristics
  * More than 4 weeks since prior and no concurrent medications that are known to inhibit the CYP2D6 system
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-03-16 (Actual); Primary Completion 2014-05-12 (Actual); Study Completion 2014-05-27 (Actual)

PRIMARY OUTCOMES:
Percent change in plasma concentrations of 4-hydroxy tamoxifen and of endoxifen after ≥ 8 weeks of concurrent administration of tamoxifen citrate and a CYP2D6 inhibitor | Between 8-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, MD, Study Chair — Mayo Clinic
Locations (6):
- United States (6):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Virginia Cancer Specialists PC-Arlington, Arlington, Virginia

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials